CLINICAL TRIAL: NCT02769780
Title: A Web-based Observational Study of Patient-reported Outcomes in Adults With Narcolepsy
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Invitae Corporation (Industry); Wake Up Narcolepsy (Unknown); Narcolepsy Network (Unknown); ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: Nexus Narcolepsy Registry
Record Dates: First submitted 2016-03-09; First posted 2016-05-12 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Nexus is a collaboration between academic institutions, advocacy and industry to answer important questions about narcolepsy. It is a web-based observational study of patient-reported outcomes in adult patients with narcolepsy, with follow-up every six months.

Nexus website: www.narcolepsyregistry.com

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with narcolepsy by a doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with narcolepsy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Descriptive epidemiology of type 1 and type 2 narcolepsy | Participants complete a survey every 6 months for 3 years after enrollment
  Assessments include disease/diagnosis characteristics, disease/symptom characteristics, health-related quality of life (HRQoL), functioning, work productivity, resource utilization, and comorbidity burden at the time of enrollment and their progression through the course of the study

SECONDARY OUTCOMES:
Medication utilization and treatment outcomes for type 1 and type 2 narcolepsy | Participants complete a survey every 6 months for 3 years after enrollment
  Assessments include: Medication use, non-pharmacologic disease management, symptom relief, quality of life (QoL), functionality and productivity associated with varying treatment regimens at baseline and their change throughout the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Hyman, PhD, Study Director — Jazz Pharmaceuticals; JeanPierre Coaquira, MPH, Principal Investigator — Jazz Pharmaceuticals
Locations (1):
- Jazz Pharmaceuticals, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Thorpy MJ, Ohayon MM, Carls G, Black J, Pasta DJ, Hyman DL, Villa KF. Assessing the impact of sodium oxybate treatment on functioning, productivity, and health-related quality of life in patients with narcolepsy: findings from the Nexus Narcolepsy Registry (waves 1-4). Sleep Med. 2021 Aug;84:380-388. doi: 10.1016/j.sleep.2021.06.010. Epub 2021 Jun 19. PMID 34247126